CLINICAL TRIAL: NCT06880978
Title: Mini-Crush Or Controlled Balloon-Crush For True Coronary Bifurcation Lesions
Status: Recruiting | Type: Observational
Sponsor: Istanbul Mehmet Akif Ersoy Educational and Training Hospital (Other Government)
Collaborators: Istanbul Medipol University Hospital (Other); Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other); Başakşehir Çam & Sakura City Hospital (Other Government); Sisli Hamidiye Etfal Training and Research Hospital (Other); Ankara Etlik City Hospital (Other Government); Ankara City Hospital Bilkent (Other); Istanbul University - Cerrahpasa (Other); Trakya University (Other); Cigli Regional Training Hospital (Other); Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government); İstanbul Bağcılar Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Ahmet Guner, Principal Investigator, Istanbul Mehmet Akif Ersoy Educational and Training Hospital
Other Study IDs: 2025.02-25
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Coronary Bifurcation Lesions; Death; Myocardial Infarction (MI); Stent Thrombosis; Stroke
Keywords: Coronary bifurcation; death; revascularization; stenting
MeSH Terms: conditions — Death; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mini-crush stenting Group: Stenting with mini-crush technique for true coronary bifurcation lesions
- Controlled balloon-crush Group: Stenting with controlled balloon-crush technique for true coronary bifurcation lesions

SUMMARY:
The mini-crush technique is one of the leading 2-stent techniques frequently applied by interventional cardiologists to treat complex bifurcation lesions. In the last 20 years, many technical innovations and iterations of mini-crush technique have been developed, and it maintains its popularity among invasive cardiologists. Moreover, mini-crush and double kissing-crush techniques have been compared in terms of clinical results in both left main and non-left main coronary bifurcation patient populations and no significant difference was found. However, the most important challenges of the mini-crush technique are the rewiring and advancement of a 1:1 non-compliant side-branch balloon after the main branch stent has been implanted. These challenges usually necessitate the use of a low profile balloon or additional support maneuvers (such as anchor balloon). Recently, a novel modified mini-crush-crush technique (controlled balloon-crush) has been introduced to the literature and is one of the most up-to-date crush techniques. The main advantage of this technique over the contemporary mini-crush technique is that the side branch can be easily rewired and the 1:1 size non-compliant balloon can easily pass through the crushed stent structure in the ostial part of the side branch. The basic rationale of this is that the crushing of the side branch stent is done in a more controlled manner (by slowly deflation of the side branch stent balloon) and this causes less disruption of the stent cells. This prospective observational study aims to assess the procedural and 1-year clinical outcomes of the contemporary mini-crush and controlled balloon-crush (modified mini-crush) double stenting techniques in patients with true coronary bifurcation lesions.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18
* PCI with mini-crush or controlled balloon-crush
* Complex coronary bifurcation lesion (Medina 0.1.1 and Medina 1.1.1)

Exclusion Criteria:

* Non-complex bifurcation anatomy
* Bail-out 2-stent (reverse mini-crush or reverse controlled balloon-crush)
* ST-elevation myocardial infarction
* Cardiogenic shock status
* In-stent restenosis
* A history of coronary artery bypass grafting
* Implantation of bare-metal stent
* End-stage hepatic or renal disease
* <1-year life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complex coronary bifurcation disease
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 12-months
  The primary endpoint is defined as the composite of the rates of major adverse cardiac events (MACE) (%) including cardiac death (%), target vessel myocardial infarction (%), and target lesion revascularization (%).

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebral events (MACCE) | 12-months
  The secondary endpoint (clinical) is defined as the composite of the rates of major adverse cardiac and cerebral events (MACCE) (%) including all-cause death (%), target vessel myocardial infarction (%), target lesion revascularization (%), probable or definite stent thrombosis (%), or stroke (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided